CLINICAL TRIAL: NCT02017457
Title: Sequential Administration of 5-azacytidine (AZA) and Donor Lymphocyte Infusion (DLI) for Patients With Acute Myelogenous Leukemia (AML) and Myelodysplastic Syndrome (MDS) in Relapse After Allogeneic Stem Cell Transplantation.
Brief Title: Azacytidine and Lymphocytes in Relapse of AML or MDS After Allogeneic Stem Cell Transplantation.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Carlos Graux, MD, PhD (Other)
Collaborators: Celgene Corporation (Industry); Belgian Hematological Society (Other)
Responsible Party: Sponsor-Investigator, Carlos Graux, MD, PhD, Professor, University Hospital of Mont-Godinne
Organization: University Hospital of Mont-Godinne (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BHS-TC-10
Record Dates: First submitted 2013-12-16; First posted 2013-12-20 (Estimated); Last update posted 2019-12-10 (Actual); Status verified 2019-12

CONDITIONS: Acute Myelogenous Leukemia; Myelodysplastic Syndrome
Keywords: Hematology; Acute Myelogenous Leukemia; Myelodysplasic syndrome; Allogeneic stem cell transplantation; Donor lymphocyte infusion; DLI; Azacytidine; Vidaza; Overall response rate; Relapse
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Myelodysplastic Syndromes; Recurrence | interventions — Azacitidine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Azacytidine + Donor lymphocyte infusion (Experimental): Azacytidine will be administered subcutaneously for 5 days. During the first cycle, a dose of 100mg/m2/day will be used and for the following cycles a dose of 35mg/m2/day will be administered. Each cycle will consist in 28 days. All patients will receive at least 6 cycles of Azacytidine and the total number of cycles will depend on the response to treatment.
  Donor lymphocyte infusion will be performed on day 1 of cycle 2, 4 and 6 of Azacytidine. The amount of cells infused will depend on donor origin.
  Interventions: Biological: Donor lymphocyte infusion; Drug: Azacytidine

INTERVENTIONS:
Biological: Donor lymphocyte infusion — On day 1 of cycle 2, 4 and 6 of Azacytidine, patients will be infused with donor lymphocytes (ideally on day 1 but in case of organizational problems, DLI can be administered until day 5) .
  * Patients with a sibling donor will receive:
  * 5x10exp7 CD3+/kg on day 1 of cycle 2
  * 5x10exp7 CD3+/kg on day 1 of cycle 4
  * 10x10exp7 CD3+/kg on day 1 of cycle 6
  * Patients with an unrelated donor will receive:
  * 1x10exp7 CD3+/kg on day 1 of cycle 2
  * 5x10exp7 CD3+/kg on day 1 of cycle 4
  * 10x10exp7 CD3+/kg on day 1 of cycle 6
  Other Names: DLI
Drug: Azacytidine — * Cycle 1: Subcutaneous administration of 100mg/m2/day for 5 days.
  * Cycle 2: Subcutaneous administration of 35mg/m2/day for 5 days. Cycles will be administered every 28 days.
  All patients will receive at least 6 cycles of Azacytidine except if progression requests additional disease-related treatment such as hydroxyurea or other chemotherapeutic agents. In such cases, the patient will be excluded from the study and only disease status and survival status will be reported during the 3-year follow-up period. In case of complete remission after cycle 5, 2 additional cycles will be administered after achievement of complete remission.
  In case of stable disease or partial response, Azacytidine will be continued until progression.
  In case of disease progression after cycle 6, Azacytidine will be stopped.
  Other Names: Vidaza

SUMMARY:
The present project is a multicenter, phase II trial which aims at evaluating if the administration of azacytidine (Vidaza®) combined to donor lymphocyte infusion (DLI) could improve the response rate to DLI in the population of patients with relapsed acute myeloid leukemia (AML) and myelodysplastic syndrome (MDS) after allogeneic hematopoietic stem cell transplantation.

DETAILED DESCRIPTION:
This is a prospective, multicenter, non-randomized phase II study. The aims at evaluating if the administration of azacytidine (Vidaza®) combined to donor lymphocyte infusion (DLI) could improve the response rate to DLI in the population of patients with relapsed acute myeloid leukemia (AML) and myelodysplastic syndrome (MDS) after allogeneic hematopoietic stem cell transplantation.

Because the investigators focus our interest on relapsed MDS and low marrow blast count relapsed AML, the investigators postulate that one cycle at higher doses of azacytidine given at 100 mg/m² during 5 days is enough to induce temporary disease control, as suggested by the predictive value of the immediate response rate after the first cycle described in the study of Czibere et al. Starting with cycle 2, the investigators propose to administer DLI along with azacytidine to optimise the immunomodulatory effect. Because these immunomodulatory effects have been described at low dose, the investigators postulate that 35 mg/m² given during 5 days is enough to harness a graft-versus-leukemia effect and induce durable remissions without exacerbating GvHD. DLI will be given every other cycle following an escalated-dose regimen.

The investigators have estimated a sample size of 50 patients to be recruited during 4 years with a 2-year follow-up and a 3-year long-term follow-up. The whole study will be completed within 9 years.

ELIGIBILITY:
Inclusion Criteria:

1. Patients:

   * Age ≥ 18 years
   * Be able to understand and sign informed consent
   * Fertile patients must use a reliable contraception method
2. Disease status at transplantation:

   * AML in first or subsequent complete remission (< 5% marrow blasts)
   * MDS with less than 10% marrow blasts at the time of transplantation
3. Transplantation:

   * Allogeneic transplantation using a sibling or unrelated donor with matching in 10/10 alleles (HLA-A, B, C, DRB1, DQB1) or maximum of one allele or one antigen or 1 antigen + 1 allele or 1 antigen + 1 DQB1 antigen or 2 alleles mismatches.
   * Myeloablative or reduced-intensity conditioning
   * Second transplantation is allowed
   * Donor is willing to donate lymphocytes
4. Clinical situation:

   * Cytological relapse after allo-SCT defined as the recurrence of more than 5% blasts on bone marrow aspiration (AML) or evidence of MDS
   * Immunophenotypic relapse defined as the recurrence of an abnormal phenotype on flow cytometry in bone marrow aspirate (only in case of a specific phenotype).
   * Cytogenetic or molecular relapse defined as the persistence or recurrence of a cytogenetic abnormality or molecular marker in bone marrow aspiration or peripheral blood. WT1 expression is not considered as reliable marker for relapse in this protocol but FLT3-ITD, NPM1, CEBPA, or translocation-specific markers (such as MLL-PTD, AML-ETO, CBFB-MYH11) are.
5. Immunosuppressive therapy should have been stopped before inclusion.

Exclusion Criteria:

* More than 30% marrow blasts at the time of inclusion
* Extramedullary relapse including CNS involvement
* ECOG Performance status > 2
* Active acute grade II-IV GvHD at the time of inclusion
* Active chronic GvHD requiring systemic therapy at the time of inclusion
* Uncontrolled infection
* HIV positive
* Acute or chronic heart failure (NYHA class III or IV) or symptomatic ischemic heart disease or ejection fraction < 35% or uncontrolled arrhythmia
* Severe liver failure (total bilirubin > 3 mg/dL, SGPT > 4 X upper normal limit)
* Severe pulmonary failure (corrected DLCo < 35%)
* Terminal renal failure requiring dialysis
* Severe neurological or psychiatric disorders
* Concurrent investigational drug.
* Other treatment for relapse, except for hydroxyurea but it should be stopped before inclusion in the study.
* Female who is pregnant or breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2013-12; Primary Completion 2019-11 (Actual); Study Completion 2019-11 (Actual)

PRIMARY OUTCOMES:
Response rate | Will be evaluated at day 24 of cycle 1, 3 and 5. Then every 3 months for a year after cycle 6 thereafter at 1.5 and 2 years after cycle 6
  To assess the response rate to DLI by the combination with azacytidine in the population of patients with relapsed AML and MDS after allo-SCT.

SECONDARY OUTCOMES:
Disease-free survival | 2 years after cycle 6
  Disease-free survival of patients
Overall survival | 2 years after cycle 6
  Overall survival of patients
Evaluation of the treatment Toxicity | At the beginning of each cycle and at the discretion of the investigator until cycle 6, then monthly for 6 months, thereafter every 3 months for 1.5 years
  Evaluate haematological and non-haematological toxicities and safety of the planned therapy.
Incidence and severity of GvHD | At the beginning of each cycle and at the discretion of the investigator until cycle 6, then monthly for 6 months, thereafter every 3 months for 1.5 years
  Incidence and severity of GvHD
Incidence and severity of infections | At the beginning of each cycle and at the discretion of the investigator until cycle 6, then monthly for 6 months, thereafter every 3 months for 1.5 years
  Incidence and severity of infections

OTHER OUTCOMES:
Immune reconstitution | On day 1 of each cycle until cycle 6, then every 3 months for a year and at 1.5 and 2 years after cycle 6
  Immune reconstitution (hemoglobuline in g/dL)
Immune reconstitution | On day 1 of each cycle until cycle 6, then every 3 months for a year and at 1.5 and 2 years after cycle 6
  Immune reconstitution (ANC, ALC, platelet in cells/µL)
Treg expansion | On day 1 of each cycle until cycle 6, then every 3 months for a year and at 1.5 and 2 years after cycle 6
  Treg expansion

CONTACTS AND LOCATIONS:
Overall Officials: Xavier Poiré, MD, Principal Investigator — Cliniques universitaires Saint-Luc- Université Catholique de Louvain; Carlos Graux, MD, PhD, Principal Investigator — Cliniques Universitaires Mont-Godinne
Locations (12):
- Belgium (12):
  - Ziekenhuis Netwerk Antwerpen, Antwerp
  - AZ Sint-Jan Brugge, Bruges
  - Institut Jules Bordet, Brussels
  - Universitair Ziekenhuis Antwerpen, Edegem
  - Universitair Ziekenhuis Gent, Ghent
  - Hopital de Jolimont, Haine-St-Paul
  - Universitair Ziekenhuis Brussel, Jette
  - Universitair Ziekenhuis Leuven, Leuven
  - CHU Liège, Liège
  - Hartziekenhuis Roeselare Menen, Roeselare
  - Cliniques Universitaires Saint-Luc, Woluwe-Saint-Lambert
  - CHU Mont-Godinne, Yvoir